CLINICAL TRIAL: NCT06714864
Title: An Open-Label, Two-Arm (DefenCath® vs. Institutional Standard of Care) Study to Assess Safety and Time to Catheter-related Bloodstream Infections (CRBSI) in Subjects From Birth to Less Than 18 Years of Age With Kidney Failure Receiving Hemodialysis Via a Central Venous Catheter
Brief Title: Open-Label Study to Assess Safety and Time to Catheter-related Bloodstream Infections (CRBSI) in Subjects From Birth to < 18 Years of Age
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CorMedix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEDI-LOCK
Expanded Access: NCT06707480 (Available)
Record Dates: First submitted 2024-12-02; First posted 2024-12-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections | interventions — taurolidine; Heparin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DefenCath® (Experimental)
  Interventions: Drug: (taurolidine and heparin) catheter lock solution
- Control (Active Comparator)
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: (taurolidine and heparin) catheter lock solution — for central venous catheter instillation use
  Other Names: DefenCath®
  Arms: DefenCath®
Drug: Standard of Care — Site specific standard of care
  Arms: Control

SUMMARY:
This study is a post-marketing approval requirement to assess the safety and time to Catheter-related Bloodstream Infections (CRBSI) of DefenCath in pediatric population (birth to less than 18 years of age) who are on chronic HD for kidney failure.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be < 18 years of age and must meet the following inclusion criteria:
* The investigator, or a person designated by the investigator, will obtain written informed consent from each study participant's legal guardian and the participant's assent, when applicable, before any study-specific activity is performed. All legal guardians should be fully informed, and participants should be informed to the fullest extent possible, about the study in language and terms they are able to understand.
* A legal guardian or primary caregiver must be available to help the study-site personnel ensure follow up; accompany the participant to the study site on each assessment day according to the schedule of activities (SoA) (e.g., able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures); consistently and consecutively be available to provide information on the participant during the scheduled study visits; accurately and reliably dispense study intervention as directed.
* The participant has kidney failure and undergoes chronic hemodialysis (HD) at least 2 times per week.
* The participant has an HD central venous catheter (CVC) and is placed in a jugular or subclavian vein.
* The participant has demonstrated the ability to achieve an appropriate minimum blood flow (Qb) for the participant's relative age and weight for at least 2 consecutive dialysis sessions to enable successful HD.
* The participant is likely to require the use of a CVC for at least 60 days, based on clinical assessment.
* The participant is willing to comply with specified follow-up evaluations and prescribed dialysis therapy.
* The participant is receiving adequate HD as assessed by the investigators and based on a single pool Kt/V measurement > 1.2 (within the last 40 days).
* The participant is not expected to expire within 180 days, based on clinical assessment.
* Female participants of childbearing potential:
* Must agree to abide by contraception requirements, must not be lactating, and avoid pregnancy during study participation from the first Screening visit until 30 days after the last administration of study treatment.
* Must commit to an additional method of birth control in addition to male partners agreeing to use condoms with spermicide, throughout the study including for at least 30 days after the last administration of study treatment:
* True abstinence: Refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the participant (periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable).

Combined (containing estrogen and progestogen) hormonal birth control (oral, intravaginal, injectable, or transdermal) associated with inhibition of ovulation initiated at least 30 days before dose administration.

* Progestogen only hormonal birth control (oral, injectable, or implantable) associated with inhibition of ovulation initiated at least 30 days before study dose administration.
* Bilateral tubal occlusion/ligation.
* Intrauterine device.
* Intrauterine hormone releasing system.
* Vasectomized partner.
* NOTE: If the childbearing potential changes after start of the study (e.g., a premenarchal female participant experiences menarche) or the risk of pregnancy changes (e.g., a female participant who is not heterosexually active becomes active), the participant must discuss this with the investigator, who should determine if a female participant must begin a highly effective method of contraception, or a male participant must use a condom. If reproductive status is questionable, additional evaluation should be considered.
* Male participants who are sexually active with a female partner of childbearing potential must agree to use male condoms and spermicide, even if the male participant has undergone a successful vasectomy (males with vasectomy can use condoms without spermicide), from Day 1 until at least 30 days after the last administration of study treatment.

Exclusion Criteria:

* The participant has received systemic antibiotics within the last 14 days. Topical antibiotic use is permitted.
* Visible evidence of compromised skin integrity is present at the catheter exit site or evidence of a catheter exit site infection.
* The participant has received any thrombolytic treatment (i.e., tissue plasminogen activator [tPA] - Cathflo®), not as part of the institution's standard of care for patency management, in their current catheter within 30 days of randomization.
* The fill volume of catheter lumen(s) is unknown or cannot be determined.
* The participant uses any type of antimicrobial-coated or heparin-coated catheter.
* Documented chronic bleeding diathesis, active or recurrent bleeding within 30 days prior to randomization.
* Documented history of an atrial thrombus or known hypercoagulable state.
* The participant has open, non-healing skin ulcers.
* Current requirement for systemic immunosuppression that would increase risk of infection, such as:
* High dose steroid. Low-dose steroids, such as routinely used for maintenance of organ transplants, are acceptable.
* Methotrexate dose sufficiently high to suppress white blood cells (WBC) below 5,000 cells/µL.
* Biologic immunomodulators (anti-tumour necrosis factor, anti-CD4 antibody, etc.) within 30 days.
* Azathioprine.
* Calcineurin inhibitors (dose determined by investigator).
* Sirolimus.
* An active malignancy that either in and of itself or by virtue of its treatment with chemotherapy or biologic therapy results in neutropenia, leukopenia and/or immunosuppression.
* Known allergy or absolute contraindication to taurolidine, citrate, or heparin, or a history of heparin induced thrombocytopenia (HIT).
* Unstable malignancy.
* Cirrhosis with encephalopathy.
* The participant is currently taking another medication with known systemic drug interaction with taurolidine, citrate, or heparin.
* The participant is anticipated to receive a renal transplant within 90 days (participants can be on the transplant list, but a participant with a known or anticipated transplant date within the next 90 days should be excluded).
* The participant has a clinically significant cardiac rhythm or functional disorder.
* The participant has severe hypoxemia, respiratory acidosis, asphyxia, or hypotension prior to randomization based on assessment of the investigator.
* Any other medical condition which renders the participant unable to or unlikely to complete the study, or which would interfere with optimal participation in the study or produce significant risk to the participant.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time to first clinical diagnosis of Catheter-related Bloodstream Infections (CRBSI) | Patient has been randomized and has received at least 1 instillation of the assigned lock solution, and has received confirmed diagnosis of CRBSI (up to 13 months)
  To demonstrate the effectiveness of DefenCath as a catheter lock solution (CLS) for prevention of CRBSI in pediatric participants receiving chronic hemodialysis (HD) through a central venous catheter (CVC) for the treatment of kidney failure.
Descriptive analysis characterizing the relative rates of deaths, AEs, and SAEs | Patient has been randomized and has received at least 1 instillation of the assigned lock solution, and has received confirmed diagnosis of CRBSI (up to 13 months)
  To demonstrate safety of DefenCath as a CLS in pediatric participants receiving chronic HD through a CVC for the treatment of kidney failure

SECONDARY OUTCOMES:
Time to catheter removal due to CRBSI | Patient has been randomized and has received at least 1 instillation of the assigned lock solution, and has received confirmed diagnosis of CRBSI (up to 13 months)
  To evaluate the catheter removal due to CRBSI in pediatric participants who are receiving chronic HD through a CVC for kidney failure.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Children's of Alabama/University of Alabama, Birmingham, Alabama
  - Stanford, Palo Alto, California
  - Nemours Children's Hospital - DE, Wilmington, Delaware
  - Cook Children's Health Care System, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Undecided